CLINICAL TRIAL: NCT00905112
Title: Musculoskeletal and Obstetric Management Study (MOMS)
Brief Title: Musculoskeletal and Obstetric Management Study
Acronym: MOMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Logan College of Chiropractic (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); Washington University School of Medicine (Other)
Responsible Party: Dr. Clayton Skaggs, Logan University, College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-0998; 417 (DRD); 1 R18HP07640-01-00 (Award #); R18HP07640 (Grant #); RD1012060046 (Logan IRB #)
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2009-05-20 (Estimated); Status verified 2009-05

CONDITIONS: Lower Back Pain; Pelvic Pain; Musculoskeletal Pain
Keywords: Pregnancy; Pain; Musculoskeletal manipulations; Exercise
MeSH Terms: conditions — Low Back Pain; Pelvic Pain; Musculoskeletal Pain; Pain; Motor Activity | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MOMS (Experimental): Receives manual therapy, stabilization exercise and patient education
  Interventions: Other: Manual Therapy
- STOB (Active Comparator): Receive standard obstetrical care
  Interventions: Other: Standard OB Care

INTERVENTIONS:
Other: Manual Therapy — Receives manual therapy, stabilization exercise and patient education
  Arms: MOMS
Other: Standard OB Care — Receive standard obstetrical care
  Arms: STOB

SUMMARY:
The investigators propose such a trial to compare a Musculoskeletal and Obstetric Management (MOM) program to standard obstetric care alone for lower back pain/pelvic pain (LBP/PP) during and after pregnancy.

DETAILED DESCRIPTION:
Initially patients will have a Baseline Musculoskeletal Exam (BME) at 24-28 weeks pregnancy at which point self reported tests/questionnaires will be administered as well as functional testing (see below "procedures for research") performed. At this point patients will be randomized into either Standard Obstetric Management or Musculoskeletal and Obstetric Care (MOMS) groups:

Standard Obstetric Management : All patients (both groups) will be seen for standard obstetric care typically once every month. Complicated cases may need to be seen more frequently. There is no standard obstetric care approach to LBP/PP in pregnancy, thus, patients in the standard obstetric care group will receive limited, although realistic interventions for LBP/PP. In addition, patients will attend one-on-one educational sessions on pre-natal care. The women in this group will have a minimum of 4 pre-natal care sessions. These visits will be timed to match the additional time and care given to the MOM group. The timed sessions will be compared with the MOMS group at monthly intervals to maintain treatment attention equality. Patients will have a complete medical assessment including history and physical examination administered by their obstetrical provider. As part of their intervention for LBP/PP, evaluation of lifestyle and work activities may be taken into consideration. Modification of lifestyle may be recommended including, rest and general aerobic exercise. Short-lived heat treatment (i.e. heating pad for no more than 10 minutes) is another possibility. Use of analgesia may be prescribed, including acetaminophen and NSAID preparations, or narcotics if deemed necessary by the provider. Narcotic use and centrally acting muscle relaxants are typically not encouraged, but at times maybe necessary to help control pain. For pain that is debilitating and worsening, consultation with orthopedic or neurological services may be considered.

Musculoskeletal and Obstetric Management (MOM): In addition to their standard obstetric visits, patients in this group will see the MOM team every one to two weeks depending on severity of symptoms. We have found through treating pregnancy-related pain that visits every one to two weeks is sufficient as the majority of the cases are mild to moderate presentations of non-inflammatory pain. A standard history will be taken and the patient will be assessed for musculoskeletal conditions to identify signs of serious illness, neurological deficit and/or orthopedic instability. If any of these conditions are evident, the patient will be immediately referred for specialist consultation. The patients in this MOM group will be treated with biobehavioral management, manual therapy and spinal stabilization exercise as described in detail below. The obstetric physician and chiropractic physician will have coordinated schedules at each clinic. For pain that is debilitating and worsening, consultation with orthopedic or neurological services will be considered.

Patients will be assessed at 33 weeks gestation and 3 months post-partum and research end-points collected. Please see next cell for detailed description of these functional and endurance tests as well as self reported test.

ELIGIBILITY:
Inclusion Criteria:

* Female Patients 15-45 years of age
* Pregnant - 24-28 weeks gestation
* LBP and/or PP

Exclusion Criteria:

* History of fracture, neoplasm, previous surgery of lumbar spine, pelvis, hip or femur
* Acute inflammatory or infectious disease
* Chronic pain prior to pregnancy (pain persisting for > 8 weeks prior to pregnancy)
* Mental health disorder requiring medication/treatment
* Back pain from visceral diseases
* Peripheral vascular disease and/or cardiac disease requiring medical treatment
* Severe disabling health problems
* Substance abuse
* Ongoing treatment for back pain by other health care providers
* Pending or current litigation
* Multiple birth pregnancies

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2006-10; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Quebec Task Force Disability Scale Questionnaire (QDQ) | Baseline, 33 weeks of gestation and 3 months postpartum

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) | Baseline, 33 weeks of gestation and 3 months postpartum
Personal Pain History (PPH) | Baseline, 33 weeks of gestation and 3 months postpartum
Straight Leg Raise (SLR) | Baseline, 33 weeks of gestation and 3 months postpartum
Active Straight Leg Raise (ASLR) | Baseline, 33 weeks of gestation and 3 months postpartum
Long Dorsal Ligament Test (LDLT) | Baseline, 33 weeks of gestation and 3 months postpartum
Posterior Pelvic Pain in Pregnancy Test (P4) | Baseline, 33 weeks of gestation and 3 months postpartum
Extensor Endurance Test (EET) | 3 months postpartum
Flexor Endurance Test (FET) | 3 months postpartum
Side Bridge (SB) | 3 months postpartum

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Center for Advanced Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri